CLINICAL TRIAL: NCT03215134
Title: A Novel Intervention for Self-criticism in a Primary Care Psychological Therapies Service: Feasibility Study
Brief Title: Self-Criticism Feasibility Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Collaborators: South London and Maudsley NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 17/LO/0335
Record Dates: First submitted 2017-06-06; First posted 2017-07-12 (Actual); Last update posted 2018-08-09 (Actual); Status verified 2017-12

CONDITIONS: Self-Criticism
Keywords: Improving Access to Psychological Therapies (IAPT); Primary mental health service; Compassion Focused Therapy (CFT)

STUDY DESIGN:
Intervention Model Description: uncontrolled pilot study of 1 intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Self-criticism intervention (Experimental): 6 weekly face to face therapy sessions (1st assessment an intervention session of 60 to 90 minutes; sessions 2-5 are 60 minutes each) and a 2 month follow-up telephone call of upto 30 minutes.
  Interventions: Other: Self-criticism intervention

INTERVENTIONS:
Other: Self-criticism intervention — Compassion Focused Therapy (Gilbert, 2010) adapted to focus specifically on reducing self-criticism. This intervention was originally developed for a student population (Rose, McIntyre & Rimes, submitted) and is now being evaluated in a primary mental-health service.

SUMMARY:
This uncontrolled pilot seeks to develop a novel intervention based on Compassion Focused Therapy (CFT), that reduces self-criticism and improves psychological wellbeing. The researchers aim to assess the the acceptability and feasibility of providing such an intervention within a primary mental health care service; and a preliminary indication of the the effectiveness of this intervention?

DETAILED DESCRIPTION:
The intervention is based upon recent unpublished doctoral research that developed this novel treatment within students with high levels of self-criticism. This pilot study aims to adapt the intervention for an Improving Access to Psychological Therapies (IAPT) service, a primary mental-health service in the UK.

Self-criticism is a transdiagnostic process across common mental-health disorders and is therefore, a potential target for psychological intervention. Clients at IAPT are likely to present with high levels of self-criticism. This pilot study may help develop an alternative evidence-based intervention that can be routinely offered within IAPT services.

The researchers aim to recruit 20 clients registered at Talking Therapies Southwark, experiencing a significant impact of self-criticism on their daily life, and requesting help for self-criticism. Clients that provide consent to participate in this study would receive 6 sessions of this intervention and a 2-month follow-up telephone session.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent
2. Registered with and opt into the Southwark IAPT service, Talking Therapies Southwark
3. Score at least 10 on the WSAS questionnaire regarding the impact of self-criticism on their daily life
4. Requesting help for their self-criticism.

Exclusion Criteria:

1. Not being sufficiently proficient in English to fully participate in the sessions with English-speaking therapists or process the written study materials for any reason.
2. Being unable to attend six sessions of assessment/treatment.
3. Presenting with high levels of risk requiring monitoring and assistance beyond the weekly intervention focusing on self-criticism.
4. Current serious mental health problem such as bipolar disorder, anorexia nervosa or a moderate / severe substance use disorder.
5. Cognitive impairment or psychomotor retardation of a degree that would prevent completion of the study treatment protocol with the individual. This would be based on a clinical judgement by potential referrers or by the clinician undertaking the screening assessment.
6. Currently experiencing a degree of life stress (e.g. recent bereavement) that is judged by the assessor to be likely to seriously adversely affect their ability to benefit from the intervention
7. New pharmacological interventions for psychological distress - i.e. a change of medication or dosage in the last 4 weeks.
8. Current participation in another clinical (talking therapy or drug) trial or another psychological intervention.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-05-04 (Actual); Primary Completion 2018-04-20 (Actual); Study Completion 2018-06-12 (Actual)

PRIMARY OUTCOMES:
Do clients find the intervention an acceptable treatment option | 3.5 months (from start to end of therapy, including follow-up)
  This will be assessed through anonymised written feedback
Is this intervention feasible to deliver within an IAPT service | 9 months - through recruitment until the end of therapy for the final participant.
  This will be assessed through recruitment and retention rates
Work and Social Adjustment Scale (W&SAS) adapted to reflect self-criticism | Change from baseline will be measured again at each time-point: session 1,2,3,4,5, 6; and 2 months after session 6.
  Measure of the impact of the presenting problem, in this case, self-criticism. Change is being assessed.
Self-Critical Rumination Scale (SCRS) | Change from baseline will be measured again at each time-point: session 1,2,3,4,5, 6; and 2 months after session 6.
  Measure of self-criticism. Change is being assessed.

SECONDARY OUTCOMES:
Patient Health Questionnaire (PHQ-9) | Change from baseline will be measured again at each time-point: session 1,2,3,4,5, 6; and 2 months after session 6.
  Depressive symptoms scale. Change is being assessed.
Generalised Anxiety Disorder scale (GAD-7) | Change from baseline will be measured again at each time-point: session 1,2,3,4,5, 6; and 2 months after session 6.
  Anxiety related symptoms scale. Change is being assessed.
Rosenberg Self-Esteem Scale | Change from baseline will be measured again at session 1,4,6, and 2 months after session 6.
  Measure of self-esteem. Change is being assessed.
Habitual Index of Negative Thinking | Change from baseline will be measured again at session 1,4,6, and 2 months after session 6.
  Measure of negative self-thinking. Change is being assessed.
Forms of Self-Criticising/Attacking and Self-Reassuring Scale | Change from baseline will be measured again at session 1,4,6, and 2 months after session 6.
  measure of criticism. Change is being assessed.

OTHER OUTCOMES:
Self-Compassion Scale | Change from baseline will be measured again at session 1,4,6, and 2 months after session 6.
  Process measure reflecting levels of self-compassion. Change is being assessed.
Beliefs about Emotion Scale | Change from baseline will be measured again at session 1,4,6, and 2 months after session 6.
  Process measure reflecting the acceptability of negative emotions. Change is being assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Mehul Elliott-Joshi, Principal Investigator — Institute of Psychiatry, Psychology and Neuroscience (IoPPN), Kings College London; South London and Maudsley (SLaM) NHS Foundation Trust
Locations (1):
- South London and Maudsley NHS Foundation Trust (SlaM) and Institute of Psychiatry, Psychology and Neuroscience (IoPPN), King's College London (KCL), London, United Kingdom

IPD SHARING:
Plan to Share IPD: No